CLINICAL TRIAL: NCT03345004
Title: A Phase IIb, 2-Arm, Randomized, Double-blind, Placebo-Controlled, Multicentre Study to Optimize Diamyd Therapy Administered Into Lymph Nodes Combined With Oral Vitamin D to Investigate the Impact on the Progression of Type 1 Diabetes
Brief Title: Diamyd Administered Into Lymph Nodes in Combination With Vitamin D in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diamyd Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAGNODE-2 (D/P2/17/6); 2017-001861-25 (EudraCT Number)
Record Dates: First submitted 2017-11-01; First posted 2017-11-17 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases; Metabolic Disease; Glucose Metabolism Disorders; Immune System Diseases; Endocrine System Diseases; Juvenile Diabetes; Insulin Dependent Diabetes; Autoimmune Diabetes; Vitamin D; Physiological Effects of Drugs
Keywords: Diamyd; Diabetes; Juvenile Diabetes; Diabetes Type 1; Type 1 Diabetes; Autoimmune Diabetes; Insulin Dependent Diabetes; Type 1 Diabetes Mellitus; rhGAD65; GAD65; Diabetes Mellitus; Diabetes Mellitus Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Vitamin D; Vitamins; Micronutrients; Cholecalciferol; Ergocalciferols
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases; Metabolic Diseases; Glucose Metabolism Disorders; Immune System Diseases; Endocrine System Diseases | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The study is a 2-arm, randomized, double-blind, placebo-controlled, multicenter, clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Patients will be assigned to receive i) three (3) intralymphatic injections with Recombinant human Glutamic Acid Decarboxylase adsorbed to Alhydrogel (Diamyd) on Days 30, 60, and 90 and; ii) oral vitamin D 2000 IU/daily for 4 months (from Day 1 through Day 120)
  Interventions: Biological: Diamyd; Dietary Supplement: Vitamin D
- Placebo arm (Placebo Comparator): Patients will be assigned to receive i) three (3) intralymphatic injections of Placebo for Diamyd on Days 30, 60, and 90 and; ii) oral Placebo for vitamin D once a day for 4 months (from Day 1 through Day 120)
  Interventions: Biological: Placebo for Diamyd; Dietary Supplement: Placebo for Vitamin D

INTERVENTIONS:
Biological: Diamyd — Alhydrogel®-formulated recombinant human glutamic acid decarboxylase (rhGAD65)
  Other Names: GAD-alum
  Arms: Active arm
Dietary Supplement: Vitamin D — Oil suspension of Vitamin D
  Arms: Active arm
Biological: Placebo for Diamyd — Alhydrogel® only
  Arms: Placebo arm
Dietary Supplement: Placebo for Vitamin D — Placebo oil suspension for Vitamin D
  Arms: Placebo arm

SUMMARY:
The objective of DIAGNODE-2 is to evaluate the efficacy of Diamyd compared to Placebo, upon administration directly into a lymph node in combination with an oral vitamin D/Placebo regimen, in terms of preserving endogenous insulin secretion as measured by C-peptide.

DETAILED DESCRIPTION:
The study is a 2-arm, randomized, double-blind, placebo-controlled, multicenter, clinical trial. Eligible patients will receive injections of Diamyd/placebo into an inguinal lymph gland at three occasions, with one month intervals in combination with an oral vitamin D/placebo regimen (starting 1 month ahead of injections) during 4 months. All patients will continue to receive intensive insulin treatment from their personal physicians during the whole study period. The patients will be followed in a blinded manner for a total of 15 months. All patients that have not performed the 15 months visit when the updated protocol is implemented, will be asked to participate in the Extension Study Period which includes an additional visit at month 24.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given by patients and/or patient's parent(s) or legal acceptable representative(s) (guardian(s)) according to national regulations
2. Type 1 Diabetes (T1D) according to the Amercian Diabetes Association (ADA) classification diagnosed ≤6 months at the time of screening
3. Age: ≥12 and <25 years old
4. Fasting C-peptide ≥0.12 nmol/L (0.36 ng/ml) on at least one occasion (maximum 2 tests on different days within a period of 2 weeks)
5. Positive for Glutamic Acid Decarboxylase isoform 65 (GAD65A) but < 50 000 IU/ml
6. Females must agree to avoid pregnancy and have a negative urine pregnancy test. Patients of childbearing potential must agree to use adequate contraception, until one (1) year after the last administration of Diamyd. Adequate contraception is as follows:

For females of childbearing potential:

1. oral (except low-dose gestagen (lynestrenol and norestisteron)), injectable, or implanted hormonal contraceptives
2. combined (estrogen and progestogen containing)
3. oral, intravaginal or transdermal progesterone hormonal contraception associated with inhibition of ovulation
4. intrauterine device
5. intrauterine hormone-releasing system (for example, progestin-releasing coil)
6. bilateral tubal occlusion
7. vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
8. male partner using condom
9. abstinence from heterosexual intercourse

For males of childbearing potential:

1. condom (male)
2. abstinence from heterosexual intercourse

Exclusion Criteria:

1. Previous or current treatment with immunosuppressant therapy (although topical or inhaled steroids are accepted)
2. Continuous treatment with anti-inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
3. Treatment with any oral or injected anti-diabetic medications other than insulin
4. A history of anemia or significantly abnormal hematology results at screening
5. A history of epilepsy, head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles
6. Clinically significant history of acute reaction to vaccines or other drugs in the past
7. Treatment with any vaccine, including influenza vaccine, within 4 months prior to planned first study drug dose or planned treatment with any vaccine up to 4 months after the last injection with study drug.
8. Participation in other clinical trials with a new chemical entity within the previous 3 months
9. Inability or unwillingness to comply with the provisions of this protocol
10. A history of alcohol or drug abuse
11. A significant illness other than diabetes within 2 weeks prior to first dosing
12. Known HIV or hepatitis
13. Females who are lactating or pregnant (the possibility of pregnancy must be excluded by urine βHCG on-site within 24 hours prior to the Diamyd/placebo treatment)
14. Presence of associated serious disease or condition, including active skin infections that preclude intralymphatic injection, which in the opinion of the investigator makes the patient non-eligible for the study
15. Deemed by the investigator not being able to follow instructions and/or follow the study protocol

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, MD, Prof, Principal Investigator — Universitetssjukhuset i Linköping
Locations (18):
- Czechia (2):
  - Diabetes Centre, Institute of Clinical and Experimental Medicine, Prague
  - Department of Paediatrics, University Hospital Motol, Prague
- Diabeter Rotterdam, Rotterdam, Netherlands
- Spain (9):
  - Adult and Pediatrics Endocrinology and Diabetology, Hospital Universitario Cruces, Barakaldo
  - Adult Endocrinology and Diabetology, Hospital vall D' Hebrón, Barcelona
  - Pediatrics Endocrinology and Diabetology, Hospital Vall D'Hebrón, Barcelona
  - Adult Endocrinology and Diabetology, Hospital Ramón y Cajal, Madrid
  - Adult Endocrinology and Diabetology, Hospital Carlos Haya, Málaga
  - Pediatrics Endocrinology and Diabetology, Hospital Materno-Ifantil, Málaga
  - Adult Endocrinology and Diabetology, Hospital Macarena, Seville
  - Pediatrics Endocrinology and Diabetology, Hospital Virgen del Rocío, Seville
  - Adult and Pediatrics Endocrinology and Diabetology, Hospital Miguel Servet, Zaragoza
- Sweden (6):
  - Barn- och Ungdomskliniken, Universitetssjukhuset, Linköping
  - Endokrinmedicinska kliniken. Universitetssjukhuset, Linköping
  - Barn-och Ungdomsmedicinmottagningen and Endokrinmottagningen, Skånes Universitetssjukhus, Malmo
  - Barn- och ungdomskliniken, Uddevalla Sjukhus, Uddevalla
  - Diabetesmottagningen, Uddevalla Sjukhus, Uddevalla
  - Barnmottagningen, Norrlands Universitetssjukhus, Umeå

REFERENCES:
- [Background] Ludvigsson J, Wahlberg J, Casas R. Intralymphatic Injection of Autoantigen in Type 1 Diabetes. N Engl J Med. 2017 Feb 16;376(7):697-699. doi: 10.1056/NEJMc1616343. No abstract available. PMID 28199812
- [Background] Ludvigsson J, Tavira B, Casas R. More on Intralymphatic Injection of Autoantigen in Type 1 Diabetes. N Engl J Med. 2017 Jul 27;377(4):403-5. doi: 10.1056/NEJMc1703468. No abstract available. PMID 28745988
- [Derived] Puente-Marin S, Dietrich F, Achenbach P, Barcenilla H, Ludvigsson J, Casas R. Intralymphatic glutamic acid decarboxylase administration in type 1 diabetes patients induced a distinctive early immune response in patients with DR3DQ2 haplotype. Front Immunol. 2023 Feb 2;14:1112570. doi: 10.3389/fimmu.2023.1112570. eCollection 2023. PMID 36817467
- [Derived] Nowak C, Lind M, Sumnik Z, Pelikanova T, Nattero-Chavez L, Lundberg E, Rica I, Martinez-Brocca MA, Ruiz de Adana M, Wahlberg J, Hanas R, Hernandez C, Clemente-Leon M, Gomez-Gila A, Ferrer Lozano M, Sas T, Pruhova S, Dietrich F, Puente-Marin S, Hannelius U, Casas R, Ludvigsson J. Intralymphatic GAD-Alum (Diamyd(R)) Improves Glycemic Control in Type 1 Diabetes With HLA DR3-DQ2. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2644-2651. doi: 10.1210/clinem/dgac343. PMID 35665810
- [Derived] Ludvigsson J, Sumnik Z, Pelikanova T, Nattero Chavez L, Lundberg E, Rica I, Martinez-Brocca MA, Ruiz de Adana M, Wahlberg J, Katsarou A, Hanas R, Hernandez C, Clemente Leon M, Gomez-Gila A, Lind M, Lozano MF, Sas T, Samuelsson U, Pruhova S, Dietrich F, Puente Marin S, Nordlund A, Hannelius U, Casas R. Intralymphatic Glutamic Acid Decarboxylase With Vitamin D Supplementation in Recent-Onset Type 1 Diabetes: A Double-Blind, Randomized, Placebo-Controlled Phase IIb Trial. Diabetes Care. 2021 Jul;44(7):1604-1612. doi: 10.2337/dc21-0318. Epub 2021 May 21. PMID 34021020
- See also: Information regarding the clinical trial — http://www.diagnode-2.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Arm: Patients will be assigned to receive i) three (3) intralymphatic injections with 4µg recombinant human Glutamic Acid Decarboxylase adsorbed to Alhydrogel (Diamyd) on Days 30, 60, and 90 and; ii) oral vitamin D 2000 IU/daily for 4 months (from Day 1 through Day 120)
Period: Overall Study
Arm/Group | Active Arm | Placebo Arm
Started | 57 | 52
Haplotype DR3-DQ2 Population Month 15 | 29 | 19
Completed | 56 | 51
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Arm: Patients will be assigned to receive i) three (3) intralymphatic injections with 4µg Diamyd (GAD-alum) on Days 30, 60, and 90 and; ii) oral vitamin D 2000 IU/daily for 4 months (from Day 1 through Day 120)
  GAD-alum: Alhydrogel®-formulated recombinant human glutamic acid decarboxylase (rhGAD)
  Vitamin D: Oil suspension of Vitamin D
- Placebo Arm: Patients will be assigned to receive i) three (3) intralymphatic injections of Placebo for Diamyd (GAD-alum) on Days 30, 60, and 90 and; ii) oral Placebo for vitamin D once a day for 4 months (from Day 1 through Day 120)
  Placebo for Diamyd (GAD-alum): Alhydrogel® only
  Placebo for Vitamin D: Placebo oil suspension for Vitamin D
- Total: Total of all reporting groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 57 | 52 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (3.8) | 16.6 (4.3) | 16.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 36 | 26 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Stimulated C-peptide During a MMTT
Description: Change in C-peptide between Baseline and 15 Months. C-peptide was measured by Area Under the Curve [AUC] at 0-120 min during a Mixed Meal Tolerance Test (MMTT) and divided by 120 min. The results are given as the ratio (back-transformed from log-scale) between 15 Months and Baseline as predicted by the MMRM (Mixed Model Repeated Measures) model.
Time Frame: Baseline and 15 months
Population: Full analysis set, consist of all randomized patients who have received at least one dose of study medication and have at least one postbaseline assessment and corresponding baseline measurement of any efficacy variable. 1 patient in the active arm and 4 patients in the placebo arm were excluded due to lack of primary efficacy data at Visit 7.
Measure: Mean (Standard Deviation); unit: Unitless back-transformed from log-scale
Groups:
- Active Arm; Active (HLA DR3-DQ2): Patients will be assigned to receive i) three (3) intralymphatic injections with 4µg Diamyd (GAD-alum) on Days 30, 60, and 90 and; ii) oral vitamin D 2000 IU/daily for 4 months (from Day 1 through Day 120)
- Placebo Arm; Placebo (HLA DR3-DQ2): Patients will be assigned to receive i) three (3) intralymphatic injections of Placebo for Diamyd (GAD-alum) on Days 30, 60, and 90 and; ii) oral Placebo for vitamin D once a day for 4 months (from Day 1 through Day 120)
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 55 | 48 | 29 | 17
Unitless back-transformed from log-scale | 0.551 (1.715) | 0.506 (2.163) | 0.663 (1.511) | 0.425 (2.436)
Statistical Analysis 1: Comparison: Active Arm vs Placebo Arm; Test type: Superiority; p = 0.5009, Mixed Models Analysis; Estimated ratio = 1.091, 95% CI 2-sided [0.845 to 1.408]
Statistical Analysis 2: Comparison: Active (HLA DR3-DQ2) vs Placebo (HLA DR3-DQ2); Test type: Superiority; p = 0.0078, Mixed Models Analysis; Estimated ratio = 1.557, 95% CI 2-sided [1.126 to 2.153]

2. Secondary Outcome: Change in IDAA1c
Description: Change in insulin-dose-adjusted HbA1c (IDAA1c)
Time Frame: Baseline and 15 months
Population: Full analysis set, consist of all randomized patients who have received at least one dose of study medication and have at least one postbaseline assessment and corresponding baseline measurement of any efficacy variable. Patients with missing data are excluded.
Measure: Mean (Standard Deviation); unit: Percent of glycated hemoglobin
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 51 | 44 | 28 | 15
Percent of glycated hemoglobin | 0.757 (1.851) | 0.377 (2.183) | 0.663 (1.627) | 0.667 (2.788)

3. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c (mmol/mol)
Time Frame: Baseline and 15 months
Population: Full analysis set, consist of all randomized patients who have received at least one dose of study medication and have at least one postbaseline assessment and corresponding baseline measurement of any efficacy variable.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 56 | 51 | 29 | 18
mmol/mol | 0.53 (14.57) | 1.04 (15.87) | 0.87 (14.34) | -0.98 (18.75)

4. Secondary Outcome: Change in Insulin Consumption
Description: Change in daily exogenous insulin consumption (IU)
Time Frame: Baseline and 15 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/kg/24h
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 51 | 44 | 28 | 15
IU/kg/24h | 0.183 (0.285) | 0.094 (0.342) | 0.143 (0.196) | 0.153 (0.399)

5. Secondary Outcome: Change in Glycemic Variability/Fluctuations
Description: Change in glycemic variability/fluctuations (evaluated from data from continuous glucose monitoring FreeStyle LibrePro, FGM) over 14 day period.
Time Frame: Screening and 15 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: glycemic variability/fluctuation per day
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 49 | 39 | 25 | 12
glycemic variability/fluctuation per day
  70-180 mg/dL (hours) | -2.479 (4.638) | -2.451 (4.012) | -1.724 (3.346) | -3.920 (4.090)
  50-70 mg/dL (hours) | -0.035 (2.416) | 0.197 (1.961) | 0.034 (2.992) | 0.581 (1.057)
  <50 mg/dL (minutes) | 15.7 (46.7) | 9.0 (88.4) | 16.7 (59.3) | 48.1 (107.0)

6. Secondary Outcome: Percentage of Patients With IDAA1c ≤ 9
Description: Percentage of patients with IDAA1c ≤ 9
Time Frame: 15 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent of patients
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 51 | 44 | 28 | 15
Percent of patients | 62.7 [48.1 to 75.9] | 61.4 [45.5 to 75.6] | 78.6 [59.0 to 91.7] | 40.0 [16.3 to 67.7]

7. Secondary Outcome: Stimulated Maximum C-peptide Above 0.2 Nmol/L
Description: Percentage of patients with a stimulated maximum C-peptide level above 0.2 nmol/L (0.6 ng/ml)
Time Frame: 15 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent of patients
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 55 | 49 | 29 | 17
Percent of patients | 92.7 [82.4 to 98.0] | 75.7 [61.1 to 86.7] | 96.6 [82.2 to 99.9] | 70.6 [44.0 to 89.7]

8. Secondary Outcome: Stimulated C-peptide Above 0.2 Nmol/L at 90 Min
Description: Percentage of patients with a stimulated 90min C-peptide level above 0.2 nmol/L (0.6 ng/ml)
Time Frame: 15 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent of patients
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 55 | 49 | 29 | 17
Percent of patients | 87.3 [75.5 to 94.7] | 71.4 [56.7 to 83.4] | 96.6 [82.2 to 99.9] | 64.7 [38.3 to 85.8]

9. Secondary Outcome: Number of Hypoglycemias
Description: Number of self-reported episodes of severe hypoglycemia (Severe hypoglycemia defined as needing help from others and/or seizures and/or unconscious) (counts)
Time Frame: Baseline and 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at leastone injection.
Measure: Number; unit: Episodes
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 57 | 52 | 29 | 19
Episodes | 0 | 6 | 0 | 0

10. Secondary Outcome: Number of Patients Having at Least 1 Severe Hypoglycemic Event
Description: Number of patients having at least 1 severe hypoglycemic event (counts)
Time Frame: Baseline and 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at leastone injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 57 | 52 | 29 | 19
Participants | 0 | 1 | 0 | 0

11. Secondary Outcome: Change in Maximum C-peptide
Description: Change in maximum C-peptide during MMTT (nmol/L)
Time Frame: Baseline and 15 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 55 | 49 | 29 | 17
nmol/L | -0.350 (0.463) | -0.300 (0.350) | -0.257 (0.400) | -0.277 (0.349)

12. Secondary Outcome: Change in Fasting C-peptide
Description: Change in Fasting C-peptide (nmol/L)
Time Frame: Baseline and 15 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 55 | 49 | 29 | 17
nmol/L | -0.115 (0.148) | -0.106 (0.169) | -0.081 (0.100) | -0.095 (0.190)

13. Secondary Outcome: C-peptide Levels During a MMTT
Description: C-peptide measured at 30, 60, 90, and 120 minutes during MMTT (nmol/L) at 15 months
Time Frame: 15 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Active Arm | Placebo Arm | Active (HLA DR3-DQ2) | Placebo (HLA DR3-DQ2)
Number analyzed (Participants) | 55 | 49 | 29 | 19
nmol/L
  30 min | 0.376 (0.295) | 0.374 (0.330) | 0.659 (0.352) | 0.580 (0.282)
  60 min | 0.536 (0.383) | 0.495 (0.411) | 0.911 (0.393) | 0.715 (0.308)
  90 min | 0.645 (0.495) | 0.562 (0.438) | 1.016 (0.415) | 0.717 (0.318)
  120 min | 0.691 (0.542) | 0.590 (0.444) | 1.065 (0.430) | 0.728 (0.317)

14. Secondary Outcome: Change in Body Weight
Description: Change in body weight (kg)
Time Frame: Baseline and 15 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 56 | 51
Kg | 4.3 (5.0) | 5.6 (5.4)

15. Secondary Outcome: Injection Site Reactions
Description: Injection site reactions
Time Frame: 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at leastone injection.
Measure: Number; unit: number of episodes
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 57 | 52
number of episodes | 10 | 3

16. Secondary Outcome: Number of Clinically Significant Abnormal Results From Laboratory Measurements (Haematology and Clinical Chemistry) and Urinalysis.
Description: Number of clinically significant abnormal results from laboratory measurements (haematology and clinical chemistry) and urinalysis. (counts)
Time Frame: 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at least one injection.
Measure: Number; unit: number of significant abnormal results
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 57 | 52
number of significant abnormal results | 11 | 3

17. Secondary Outcome: Number of Clinically Significant Abnormal Results From Physical and Neurological Examinations
Description: Physical examination (general appearance including skin, mouth, throat, cardiovascular, abdomen, lymphatic glands, and neurological/musculoskeletal [including reflexes]).
  Standardised clinical neurological examination including extremity reflexes, Romberg, Walk on a line, 2 meters, Standing on 1 leg, left and right, 15 seconds per leg, Finger-nose, Mimic, Babinski reflex.
  The outcome of the assessments was recored as "normal" or "abnormal"
Time Frame: 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at leastone injection.
Measure: Number; unit: Clinically significant abnormal results
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 57 | 52
Clinically significant abnormal results
  Physical examination | 15 | 9
  Neurological examination | 4 | 0

18. Secondary Outcome: GAD65A Titer
Description: GAD65A titer (IU/ml)
Time Frame: Baseline and 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at leastone injection.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 57 | 52
IU/mL
  Baseline | 731.3 (2302.9) | 627.3 (1829.9)
  Month 15 | 19941.2 (23083.6) | 476.7 (1527.7)

19. Secondary Outcome: Number of Clinically Significant Abnormal Results in Vital Signs
Description: Vital signs (blood pressure) (mmHg)
Time Frame: 15 months
Population: Safety Analysis Set, consist of all randomized patients who received at leastone injection.
Measure: Number; unit: Clinically significant abnormal results
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 57 | 52
Clinically significant abnormal results
  Systolic blood pressure | 0 | 0
  Diastolic blood pressure | 0 | 0

20. Secondary Outcome: Change in Quality of Life (QoL)
Description: Change in QoL as measured by the standardised measure of health questionnaire EQ-5D-5L between baseline and Month 15. The EQ-5D-5L is based on 5 questions rated at 5 levels indicating from no problem (level 1) to extreme problems (level 5) regarding current state of mobility, self-care, activity, pain and anxiety. The outcome is presented as a weighted index value, where 1 is the best possible health and 0 represents being dead.
Time Frame: Baseline and 15 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Index value
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 48 | 47
Index value
  Baseline | 1.000 [0.922 to 1.000] | 1.000 [0.919 to 1.000]
  Month 15 | 1.000 [0.919 to 1.000] | 1.000 [1.000 to 1.000]

21. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI (kg/m2)
Time Frame: Baseline and 15 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 56 | 51
kg/m2 | 0.8 (1.4) | 1.3 (1.6)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events, from start of Diamyd/Placebo treatment until Month 24.
Arm/Group | Active Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/57 | 3/52
Other Adverse Events (participants affected / at risk) | 18/57 | 12/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=57) | Placebo Arm (N=52)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes Mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=57) | Placebo Arm (N=52)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (13) | 10 (17)
Viral infection (Infections and infestations) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03345004/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT03345004/SAP_001.pdf